CLINICAL TRIAL: NCT00125398
Title: A Phase II, Randomized, Open-Label Study to Examine the Safety and Efficacy of GPI 15715 for Sedation of Patients Requiring Intubation and Mechanical Ventilation in the Intensive Care Unit Setting
Brief Title: GPI 15715 For Sedation in the Intensive Care Unit (ICU) Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3000-0413; GPI 3000-0413; Sedation in an ICU Setting
Record Dates: First submitted 2005-07-28; First posted 2005-08-01 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Postoperative Sedation; Intubation; Respiration, Artificial
Keywords: AQUAVAN; GPI 15715; ICU; Sedation
MeSH Terms: conditions — Respiratory Aspiration | interventions — fospropofol

INTERVENTIONS:
Drug: AQUAVAN (fospropofol disodium; GPI 15715 )

SUMMARY:
Patients who are in the intensive care unit after surgery and require mechanical breathing support (intubation and ventilation) usually require sedation to avoid agitation and excessive stress responses. Short-acting sedatives such as midazolam and propofol are the drugs typically used for this. Propofol provides for fast sedation and fast recovery from sedation. Midazolam is slower to sedation and slower for recovery, but may provide some advantages over propofol, such as a lower incidence of hypotension (low blood pressure). This study will look at propofol compared to a product with fast sedation and recovery like that of propofol but with less of a chance for hypotension like with midazolam. Patients will be treated with the product for up to 8 hours and then will be monitored for 8 hours following treatment.

DETAILED DESCRIPTION:
Patients who are intubated and ventilated and will require up to 8 hours of sedation in the ICU are eligible for participation in this study. Patients will be randomized to receive 1 of 3 treatments. One treatment is standard of care, a propofol infusion. The other two treatment arms are infusions of GPI 15715 (AQUAVAN), one with a bolus and one without.

Patients will be treated for up to 8 hours and monitored for eight hours post treatment. If there are signs of agitation during the up to 8 hour treatment period, the infusion of the sedative medicine will be increased according to protocol.

Blood samples will be obtained periodically during the course of the study for safety evaluation and pharmacokinetic assessments. When the patient is ready for extubation or the end of the 8 hour study period has been reached, the infusion of the sedative agent will be discontinued and the patient will be monitored for 8 hours post treatment.

Guilford Pharmaceuticals was acquired by MGI PHARMA on October 3, 2005.

ELIGIBILITY:
Inclusion Criteria:

1. Require 2 to 8 hours of intubation and mechanical ventilation following elective surgery
2. American Society of Anesthesiologists (ASA) status of I-IV

Exclusion Criteria:

1. Requires emergency agency
2. Requires neuromuscular blockers during sedation
3. Requires use of epidural drug administration during sedation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-07; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of infusions

SECONDARY OUTCOMES:
Percentage of patients requiring rescue medications
Evaluation of the onset of effect
Evaluation of satisfaction with sedation
Determination of pharmacokinetic (PK) levels of GPI 15715 in blood

CONTACTS AND LOCATIONS:
Overall Officials: James Jones, MD, PharmD, Study Director — Eisai Inc.
Locations (17):
- United States (17):
  - St. Mary's Hospital, Rogers, Arizona
  - Jackson Memorial Hospital, Miami, Florida
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Central Maine Pulmonary Associates, Auburn, Maine
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Cooper University Hospital, Camden, New Jersey
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York University School of Medicine, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Department of Veterans Affairs, North Texas Health Care System, Dallas, Texas

REFERENCES:
- [Derived] Candiotti KA, Gan TJ, Young C, Bekker A, Sum-Ping ST, Kahn R, Lebowitz P, Littman JJ. A randomized, open-label study of the safety and tolerability of fospropofol for patients requiring intubation and mechanical ventilation in the intensive care unit. Anesth Analg. 2011 Sep;113(3):550-6. doi: 10.1213/ANE.0b013e31821d7faf. Epub 2011 May 19. PMID 21596879